CLINICAL TRIAL: NCT06717763
Title: Surgery Following Immune Checkpoint Inhibitions for Controlled Disease in Recurrent or Metastatic dMMR/MSI-H Colorectal Cancer
Status: Completed | Type: Observational
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Pei-Rong Ding, MD, Ph D, Sun Yat-sen University
Other Study IDs: B2020-064-Y01
Record Dates: First submitted 2024-12-01; First posted 2024-12-05 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Surgical resection for residual lesions could significantly improve the prognosis in metastatic colorectal cancers (CRCs) after systemic treatments, yet the necessity of resecting residual lesions after immune checkpoint inhibitions (ICIs) remains controversial in mismatch repair-deficient (dMMR) or microsatellite instability-high (MSI-H) diseases. We retrospectively enrolled recurrent or metastatic dMMR/MSI-H CRCs who received surgerys from Sun Yat-sen University Cancer Center. Patients without disease progression after at least 2 cycles of ICIs were included. Demographic and clinicopathological data were collected and analyzed. Relapse-free survival (RFS) after surgery were analyzed.

ELIGIBILITY:
Inclusion Criteria:

1. pathologically confirmed CRC with measurable disease per Response Evaluation Criteria in Solid Tumors (RECIST, version 1.1)20;
2. definite pathological or radiological evidence of recurrent or distant metastasis;
3. received at least 2 courses of ICIs;
4. confirmed as dMMR by immunohistochemical method or MSI-H by polymerase chain reaction or next-generation sequencing;
5. receiving therapeutic surgical treatment for residual lesions or tumor sites and achieving no evidence of disease (NED) ;
6. no progression within the duration of preoperative ICIs

Exclusion Criteria:

-

Ages: 16 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The patients with recurrent or metastatic dMMR/MSI-H CRC who received PD-1 inhibition-based ICIs and subsequently underwent surgery from January 1, 2017 to July 1, 2023 at Sun Yat-sen University Cancer Center were entrolled.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Disease-free Survival | up to 5 years
  defined as the time from randomization to the first appearance of one of the following: primary tumor recurrence, or death without cancer event; or censored at date of last follow-up
Overall Survival | up to 5 years
  defined as the time from randomization to death from any cause. Participants who were alive or lost to follow-up at the time of the analysis were censored at the date they were last known to be alive

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University, Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No